CLINICAL TRIAL: NCT03379480
Title: Examination of Therapeutic Efficacy and Potential Mechanisms of Yoga Treatment in Schizophrenia
Brief Title: Study on Examination of Therapeutic Efficacy and Potential Mechanisms of Yoga Treatment in Schizophrenia
Acronym: SATYAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Collaborators: SCARF (Schizophrenia Research Foundation ,India) Schizophrenia (Unknown)
Responsible Party: Principal Investigator, Dr Naren P Rao, Associate Professor ,Department of Psychiatry, NIMHANS, National Institute of Mental Health and Neuro Sciences, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DST/002/208/2016/00892
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Yoga; fMRI
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga arm (Active Comparator): Patients with Schizophrenia will undergo 12 sessions of yoga. According to randomization one group of patients will start yoga immediately after recruitment ,whereas another group will go into wait list for 12 weeks after which they will also undergo Yoga treatment.
  Interventions: Behavioral: Yoga arm
- Control arm (No Intervention): Healthy volunteers who will not receive yoga.

INTERVENTIONS:
Behavioral: Yoga arm — Yoga module developed for patients with Schizophrenia
  Arms: Yoga arm

SUMMARY:
The aim of this study is to examine whether yoga is efficacious as an add-on treatment for negative symptoms of schizophrenia in a randomized multi-centric trial and also to examine functional brain changes associated with self-reflection after treatment with yoga.

ELIGIBILITY:
Inclusion Criteria:

Schizophrenia Subject

1. ICD (International Classification of Diseases) 10 diagnosis of schizophrenia
2. capacity to provide informed consent, as evaluated by the MacArthur Competence Assessment Tool for Clinical Research
3. no other current comorbid axis I diagnosis (except nicotine abuse/dependence) and no general impaired intellectual functioning

Healthy volunteers:

1. Males and females between 18 and 45 years
2. Capacity to provide informed consent
3. absence of past or present psychiatric illnesses including substance abuse 4) no general impaired intellectual functioning (MMSE above24)

Exclusion Criteria:

1. Other current comorbid axis I diagnosis (except nicotine abuse/dependence) and general impaired intellectual functioning
2. History of alcohol or substance abuse or dependence in the last 12 months (with the exception of nicotine)
3. Any Contraindication to MRI like metal implants or paramagnetic objects within the body or claustrophobia (only for patients undergoing fMRI at NIMHANS)
4. Past history of head injury resulting in loss of consciousness or neurosurgery
5. Concomitant severe medical conditions
6. Change in dose of antipsychotic medication or Electroconvulsive therapy in the past 6weeks
7. Pregnant or lactating -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Improvement in negative symptoms in patients with schizophrenia | At the end of 12 weeks of yoga
  Schizophrenia patients receiving yoga as add-on treatment will have significant improvement in negative symptoms after yoga therapy compared to those in the wait-list group as reflected by a greater decrease in Scale for Assessment of negative symptoms score. This scale measures negative symptoms on a 25 item, 6-point scale. Items are listed under the five domains of affective blunting, alogia, avolition/apathy, anhedonia/asociality, and attention. A higher score indicates greater severity.

SECONDARY OUTCOMES:
fMRI changes | At the end of 12weeks
  Schizophrenia patients receiving yoga will have higher activation in Medial prefrontal cortex after yoga therapy compared to baseline and compared to those in the wait-list group at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Naren P Rao, MD, Principal Investigator — National Institute of Mental Health and Neuro Sciences, India
Locations (1):
- National Institute of Mental Health and Neurosciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Undecided